CLINICAL TRIAL: NCT04365140
Title: Alteration of the microRNA-126 Expression: a Possible Mechanism in Allergic Contact Dermatitis to Nickel
Brief Title: MicroRNA-126 and Its Target VCAM-1Dermatitis to Nickel
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Adjunt professor, Universidad Autonoma de San Luis Potosí
Other Study IDs: ACDm126
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Allergic Contact Dermatitis
Keywords: allergic contact dermatitis; nickel; microRNAs; VCAM-1
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — skin biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive ACD to nickel: Patients with positive epicutaneous patch test to nickel
- negative ACD to nickel: Patients with negative epicutaneous patch test to nickel

SUMMARY:
Background. Allergic Contact Dermatitis (ACD) is an inflammatory skin disease mediated by direct contact with allergens as nickel, the most common allergen, that may be related with epigenetic changes.

Objective. Evaluate the miR-126 expression and its target VCAM-1, in the skin of patients with ACD to nickel.

Methods. Fifteen patients with positive patch test to nickel were included, and the expression of miR-126 and VCAM-1 was evaluated by RT-qPCR.

DETAILED DESCRIPTION:
Patients that went to the dermatology and outpatient department of the Central Hospital "Dr. Ignacio Morones Prieto ", with a suspected diagnosis of nickel allergic contact dermatitis, were invited to participate in this study. Later, the objective and methodology of the study were explained to them, as well as the advantages of participating and the possible undesirable effects. All patients signed the informed consent previous perfom the medical history. After, the epicutaneous patch test was performed, and patients were divided according to the result them. Finally, under local anesthesia, two 3-mm punch biopsies, from lesional (positive parch test site) and adjacent non lesional skin, 10 cm apart, were performed. Tissues for reverse transcriptase real-time polymerase chain reaction (RT-qPCR) analyses were stored frozen in sterile tubes at 80ºC until processing

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Epicutaneous Patch Test positive to Nickel
* without previous treatment within the previous 4 weeks

Exclusion Criteria:

* Pregnancy
* nursing
* menopause
* consumption of any type of drugs (including anti-inflammatories and hormonal treatments) within the previous 2 months
* coexistence of other dermatoses conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female and male patients with allergic contact dermatitis for more than one year
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Expression of miR-126 | 9 months
  Relative expression of the miR-126 on skin biopsies from ACD patients

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Castanedo-Cazares, MD, Principal Investigator — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martins LE, Reis VM. Immunopathology of allergic contact dermatitis. An Bras Dermatol. 2011 May-Jun;86(3):419-33. doi: 10.1590/s0365-05962011000300001. English, Portuguese. PMID 21738956
- [Background] Ahlstrom MG, Thyssen JP, Wennervaldt M, Menne T, Johansen JD. Nickel allergy and allergic contact dermatitis: A clinical review of immunology, epidemiology, exposure, and treatment. Contact Dermatitis. 2019 Oct;81(4):227-241. doi: 10.1111/cod.13327. Epub 2019 Jul 9. PMID 31140194
- [Background] Cerutti C, Edwards LJ, de Vries HE, Sharrack B, Male DK, Romero IA. MiR-126 and miR-126* regulate shear-resistant firm leukocyte adhesion to human brain endothelium. Sci Rep. 2017 Mar 30;7:45284. doi: 10.1038/srep45284. PMID 28358058